CLINICAL TRIAL: NCT05211440
Title: A Randomized, Double-blind, Placebo-Controlled, Crossover Study to Investigate the Effects of Microbial Enzyme Supplementation on Postprandial Nutrient Levels and Gastrointestinal Symptoms in Healthy Middle-Aged and Older Adults
Brief Title: Microbial Enzyme Impact on Postprandial Nutrient Levels and Gastrointestinal Symptoms in Healthy Adults
Acronym: BIO-3003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: BIO-CAT, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 22237
Record Dates: First submitted 2021-11-02; First posted 2022-01-27 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Digestive Health; Gastrointestinal Health
Keywords: Enzyme; Digestion; Protease; Amylase; Lipase
MeSH Terms: interventions — Meals

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplement and placebo supplements will be provided to the clinic in blindly coded containers. The code was generated by parties not responsible for data collection, analysis, or interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Maltodextrin) (Placebo Comparator): Subjects will be directed to consume 1 placebo capsule containing maltodextrin, twice daily, for 21 days.
  Interventions: Dietary Supplement: Placebo + Meal
- BC-006 (Experimental): Subjects will be directed to consume 1 capsule containing BC-006, twice daily, for 21 days.
  Interventions: Dietary Supplement: BC-006 + Meal

INTERVENTIONS:
Dietary Supplement: Placebo + Meal — Subjects will be directed to consume 1 placebo capsule containing maltodextrin, twice daily, for 21 days. Subjects will be directed to consume the capsules with their two largest meals, in between the third and second bites of food. During the MMTT, a placebo capsule will be consumed with a standardized test meal containing chicken, peas, potatoes, and butter.
  Arms: Placebo (Maltodextrin)
Dietary Supplement: BC-006 + Meal — Subjects will be directed to consume 1 capsule containing BC-006, twice daily, for 21 days. Subjects will be directed to consume the capsules with their two largest meals, in between the third and second bites of food. During the MMTT, a BC-006 capsule will be consumed with a standardized test meal containing chicken, peas, potatoes, and butter.
  Arms: BC-006

SUMMARY:
The primary objective of this study is to investigate the acute effects of a microbial multi-enzyme mixture ("BC-006") on postprandial nutrient levels in healthy, middle-aged to older adults during a mixed meal tolerance test. Additionally, the effects of twice daily consumption of BC-006 and placebo for 3 weeks on abdominal bloating, flatulence, bowel function, and sleep quality will be measured.

DETAILED DESCRIPTION:
Digestive enzymes of the human stomach, pancreas, and small intestine, are proteins that help facilitate the breakdown of dietary macronutrients for adequate nutrient supply across tissues and organs. Protease enzymes hydrolyze dietary proteins and release the amino acid building blocks of human proteins. Lipase enzymes hydrolyze dietary fats and release monoglycerides and fatty acids which can be absorbed by enterocytes and distributed across tissues and organs for energy, immune support, and structural support. Some carbohydrase enzymes, such as a combination of amylase and glucoamylase, hydrolyze carbohydrates and release monosaccharides that fuel the grand majority of metabolism within cells of most individuals on a diet that includes carbohydrates.

Digestive function and digestive enzyme output have been shown to decline in several clinical observational studies of younger and older adults, suggesting the potential value of oral, supplemental enzymes in older adults. Supplemental enzyme preparations manufactured by fermentation of non-genetically engineered, microbial source organisms, e.g., Aspergillus spp., have been on the market for decades to support digestive health and gastrointestinal tolerance. However, clinical data in older adult subjects is lacking.

BIO-CAT's proprietary mixture of 6 microbial enzymes ("BC-006") has previously been shown in in vitro gastrointestinal simulations to promote dietary protein, fat, and carbohydrate break down better than control conditions with endogenous enzymes alone (unpublished data). BC-006 comprises a mixture of proteases, lipase, amylase, and glucoamylase. The primary objective of this clinical study is to investigate the effect of BC-006 supplementation on postprandial nutrient levels in healthy, middle-aged to older adults during a mixed meal tolerance test. Abdominal bloating, flatulence, bowel function, and sleep quality will also be measured across 3 weeks of twice daily supplementation.

This study will be a randomized, placebo-controlled, crossover design trial consisting of a preliminary virtual screen and 4 study visits (Visits 1-4). During the preliminary virtual screening, subjects will provide voluntary informed consent, subjects will undergo medical history, prior and current medication/supplement use assessments, as well as inclusion and exclusion criteria assessments. At Visit 1, subjects will arrive at the clinic in a fasting state. Height, body weight, and vital signs will be measured and BMI will be calculated from a dual-energy X-ray absorptiometry (DEXA) scan. A blood sample will be collected for rapid fasting blood glucose analysis. Upon assessment of all eligibility criteria, subjects may be enrolled and randomized to BC-006 or placebo arms. Subjects will be dispensed their assigned study product and will be instructed to consume it twice daily (2 capsules/day) with their largest meals for 21 days. Subjects will be dispensed a paper Bowel Function and Gastrointestinal Tolerance Factors Questionnaire (BF-GITFQ) to be completed daily. The BF-GITFQ contains a series of questions regarding bowel function and the presence and severity of GI symptoms occurring during the past 24 hours. Subjects will also be dispensed a paper Gastrointestinal Tolerance Questionnaire (GITQ) which contains a series of questions regarding GI symptoms occurring during the past 7 days. To assess sleep quality, subjects will be dispensed a paper Single-Item Sleep Quality Scale (SI-SQS) to be completed weekly, leading up to Visit 2.

At Visit 2, subjects will arrive at the clinic fasted and undergo clinic visit procedures (concomitant medication/supplement use, assess inclusion/exclusion criteria, body weight and vital signs measurements), and adverse event (AE) assessment. Subjects will undergo a mixed meal tolerance test (MMTT). The MMTT includes antecubital vein placement, baseline blood sample collection, provision of a standardized test meal with BC-006 or placebo, and blood sampling thereafter for 5 hours. Blood samples will be collected for analysis of free amino acids, free fatty acids, glucose, iron, and insulin. An electronic Appetite Questionnaire will also be conducted hourly during the MMTT.

Following an at least 7 day washout, subjects will return to the clinic at Visit 3 and undergo clinic visit procedures and AE assessment. Subjects will be dispensed the second study product, with instructions and questionnaires similar to the first 21 day phase of the trial. At Visit 4, subjects will arrive at the clinic fasted and undergo clinic visit procedures and AE assessment. Subjects will undergo a second MMTT with the second study product, otherwise identical to the MMTT at Visit 2.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.
2. Subject is male or female and is ≥ 40 and ≤ 75 years of age.
3. Subject has Body Mass Index (BMI) ≥ 18 but < 30 kg/m2.
4. Subject has fasting blood sugar level of 100 mg/dL or lower.
5. Subject is willing to refrain from exclusionary medications, supplements, and products throughout the study.
6. Subject is willing to follow dietary guidelines throughout the study.
7. Subject is able to follow the protocol.

Exclusion Criteria:

1. Subject states they regularly consume supplemental enzymes and are unwilling to stop at least one week prior to screening and throughout the study. Supplemental enzymes may include standalone enzyme supplements, probiotic supplements with enzymes, and any medications containing enzymes.
2. Subject states they regularly consume probiotic supplements and are unwilling to stop at least one week prior to screening and throughout the study. Supplemental probiotics may include standalone probiotic supplements, vitamins with probiotics, and any foods supplemented with probiotics.
3. Subject states they have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea, gall bladder removal).
4. Subject states they have dairy or lactose intolerance.
5. Subject states they have diabetes.
6. Subject states they have undergone bariatric surgery.
7. Subject states they have an active malignant disease, except basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix.
8. Subject states they have liver failure (decompensated chronic liver disease).
9. Subject has a stated history of a significant cardiovascular event (e.g., myocardial infarction, heart failure, or stroke) ≤ 3 months prior to screening visit.
10. Subject states they are currently diagnosed with, or has a history of severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study dietary supplement consumption or compliance with study protocol procedures in the opinion of the principal investigator or study physician.
11. Subject reports having undergone major surgery, less than 6 weeks prior to enrollment in the study, or subject has planned inpatient surgery requiring hospitalization during the study.
12. Subject states they are currently being prescribed (by primary care physician or other health professional) medication or using an over-the-counter product that in the opinion of the study physician will have an effect on food digestion or nutrient absorption during the study. Examples include prescription orlistat (Xenical) and over-the-counter orlistat (Alli).
13. Subject reports having received a COVID vaccine within 1 week of randomization or expected to receive a COVID vaccine during the study period.
14. Subject reports having previously had a positive SARS-CoV-2 test and experience symptoms for >2 months (i.e., "long-haulers").
15. Subject reports alcohol intake as average of 3 or more servings per day (a serving defined as 4 oz wine, 12 oz beer, 1 oz spirits).
16. Subject states they are pregnant or lactating or planning to become pregnant during the study.
17. Subject states they have an allergy or intolerance to any ingredient in the study product or test meal.
18. Subject is deemed unsuitable for study based upon study physician assessment.
19. Subject is taking part in another clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Total plasma essential amino acids (EAA) area under the curve (AUC) | Five hours postprandial
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined), change from baseline (BC-006 vs. placebo treatment)
Plasma EAA time-to-peak | Five hours postprandial
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined)
Plasma EAA C(MAX) | Five hours postprandial
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined)

SECONDARY OUTCOMES:
Total plasma branched chain amino acids (BCAA) AUC | Five hours postprandial
  Free leucine, isoleucine, valine (combined)
Plasma leucine AUC | Five hours postprandial
  Free leucine
Plasma total amino acids AUC | Five hours postprandial
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined)
Plasma fatty acid AUC | Five hours postprandial
  Free palmitic acid (C16:0), myristic acid (C14:0), stearic acid (C18:0), and oleic acid (C18:1n9)
Plasma glucose C(MAX) | Five hours postprandial
  Glucose (maximum)
Plasma glucose AUC | Five hours postprandial
  Glucose
Serum iron | Three hours postprandial
  Iron
Plasma insulin AUC | Five hours postprandial
  Insulin
Appetite | Five hours postprandial
  12-item Appetite Questionnaire (1 (Not at all) to 100 (Extremely))
Abdominal distension/bloating | Three weeks
  Daily, 7-item Bowel Function and Gastrointestinal Tolerance Factors Questionnaire (1 (Absent) to 4 (Severe))
Flatulence/gas | Three weeks
  Daily, 7-item Bowel Function and Gastrointestinal Tolerance Factors Questionnaire (1 (Absent) to 4 (Severe))
Individual GI symptoms other than abdominal distension/bloating and flatulence/gas | Three weeks
  Burping, cramping/pain, nausea, reflux (heartburn), rumblings (Daily, 7-item Bowel Function and Gastrointestinal Tolerance Factors Questionnaire (1 (Absent) to 4 (Severe)))
Composite score of GI symptoms (daily) | Three weeks
  Burping, cramping/pain, distension/bloating, flatulence/gas, nausea, reflux (heartburn), rumblings (Daily, 7-item Bowel Function and Gastrointestinal Tolerance Factors Questionnaire (1 (Absent) to 4 (Severe)))
Bowel function (frequency) | Three weeks
  Stool frequency (Daily, 7-item Bowel Function and Gastrointestinal Tolerance Factors Questionnaire)
Bowel function (consistency) | Three weeks
  Stool consistency (Bristol stool chart) (Daily, 7-item Bowel Function and Gastrointestinal Tolerance Factors Questionnaire (1 (Separate hard lumps, like nuts) to 7 (Watery, no solid pieces, entirely liquid)))
Bowel function (passage) | Three weeks
  Ease of stool passage (Daily, 7-item Bowel Function and Gastrointestinal Tolerance Factors Questionnaire (1 (Very easy) to 5 (Very difficult)))
Bloating | Three weeks
  Weekly, 6-item Gastrointestinal Tolerance Questionnaire (0 (No more than usual) to 2 (Much more than usual))
Gas/flatulence | Three weeks
  Weekly, 6-item Gastrointestinal Tolerance Questionnaire (0 (No more than usual) to 2 (Much more than usual))
Individual GI symptoms other than bloating and gas/flatulence | Three weeks
  Weekly, 6-item Gastrointestinal Tolerance Questionnaire (0 (No more than usual) to 2 (Much more than usual))
Composite score of GI symptoms (weekly) | Three weeks
  Nausea, bloating, gastrointestinal rumblings, gas/flatulence, abdominal pain, diarrhea (Weekly, 6-item Gastrointestinal Tolerance Questionnaire (0 (No more than usual) to 2 (Much more than usual)))
Composite sleep score | Three weeks
  Hours, ease of falling asleep, amount of times woken before waking up for day, level of refreshment (Single-Item Sleep Scale (0 (Terrible) to 10 (Excellent)))
Safety - Incidence of adverse events | Seven weeks
  Number of participants with self-reported adverse events
Safety - Incidence of any abnormal vital signs | Seven weeks
  Blood pressure, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deutz MT, Askow AT, Garvey SM, Alvarado DA, Barnes TM, Zupancic Z, Ulanov AV, Willard JW, Holscher HD, Loman BR, Burd NA. Oral multi-enzyme supplementation alters postprandial plasma nutrient concentrations after a mixed meal in healthy middle-aged and older adults: a randomized, double-blind, placebo-controlled, crossover trial. J Nutr. 2026 Feb 7:101400. doi: 10.1016/j.tjnut.2026.101400. Online ahead of print. PMID 41662956